CLINICAL TRIAL: NCT01055600
Title: A Phase IV Study Evaluating Eltrombopag Concentrations in Breast Milk of Nursing Mothers Taking Eltrombopag
Brief Title: Milk-only Lactation Study for Patients on Eltrombopag
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol opened to recruitment in Nov 2009. No potential subjects identified in 5 years; therefore, study was terminated in Jul 2014 due to lack of feasibility
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 113101
Record Dates: First submitted 2010-01-07; First posted 2010-01-25 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Thrombocytopaenia
Keywords: eltrombopag; pharmacokinetics; PROMACTA; lactation; milk-only study
MeSH Terms: conditions — Thrombocytopenia; Breast Feeding | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study (Experimental): Mothers are taking PROMACTA prescribed by their physician before entering this study. No drug will be administered as part of this study.
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — Mothers are taking PROMACTA prescribed by their physician before entering this study. No drug will be administered as part of this study.

SUMMARY:
This is a Phase IV study to evaluate eltrombopag concentrations in breast milk of nursing mothers taking marketed eltrombopag (PROMACTA®). Up to 10 subjects (mother-infant pairs) at as many as 10 study centers in the US will be enrolled. Nursing mothers who are registered with the PROMACTA Pregnancy Registry will be offered the option to participate in this trial if they continue to take commercial eltrombopag post-delivery and decide to breastfeed their infant. Information will be collected in a diary. Breast milk samples will be collected before and after infant feedings for a 24 hour period after eltrombopag dosing to evaluate the eltrombopag concentrations in the breast milk. Mothers will also be given the option to have a pharmacokinetic (PK) blood sample collected from the infant.

ELIGIBILITY:
Inclusion Criteria:

* Mother is registered with the PROMACTA Pregnancy Registry and meets all the enrollment criteria defined in the PROMACTA Pregnancy Registry study (113327).
* Mother is continuing to take eltrombopag.
* Mother has received 7 consecutive eltrombopag doses prior to the milk sample collection.
* Infant is 4 weeks to 26 weeks of age at the time of milk sampling.
* Exclusively breastfeeding mother-infant pair; either via breast or with expressed milk from the mother.
* Mother is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Infant was born with complications that could impact ability to participate in this study.
* Breastfeeding is not well established in the mother-infant pair (e.g., poor latching of the infant or low milk supply).
* Infants who are supplemented with formula or are consuming solid foods.
* Unwillingness or inability of mother to follow the procedures outlined in the protocol.
* Mother is mentally or legally incapacitated

Ages: 4 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Breast milk eltrombopag concentrations collected from nursing mothers taking eltrombopag | 24 hours

SECONDARY OUTCOMES:
AEs in infant reported during the 24 hour breast milk collection period | 24 hours
Plasma eltrombopag concentrations from infant, as data permit (optional) | 1 sample within 2 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Research Triangle Park, North Carolina, United States